#### MEDICAL RECORD

#### CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

Adult Patient or

• Parent, for Minor Patient

INSTITUTE: National Cancer Institute

STUDY NUMBER: 17-C-0116 PRINCIPAL INVESTIGATOR: Christian S. Hinrichs, M.D.

A Phase I Study of Immunotherapy with E6 T Cell Receptor T Cells for Vulvar High-

Grade Squamous Intraepithelial Lesions (HSIL)

Continuing Review Approved by the IRB on 09/24/18

Amendment Approved by the IRB on 07/09/18 (C)

Date posted to web: 10/04/18

Standard

#### INTRODUCTION

We invite you to take part in a research study at the National Institutes of Health (NIH).

First, we want you to know that:

Taking part in NIH research is entirely voluntary.

You may choose not to take part, or you may withdraw from the study at any time. In either case, you will not lose any benefits to which you are otherwise entitled. However, to receive care at the NIH, you must be taking part in a study or be under evaluation for study participation.

You may receive no benefit from taking part. The research may give us knowledge that may help people in the future.

Second, some people have personal, religious or ethical beliefs that may limit the kinds of medical or research treatments they would want to receive (such as blood transfusions). If you have such beliefs, please discuss them with your NIH doctors or research team before you agree to the study.

Now we will describe this research study. Before you decide to take part, please take as much time as you need to ask any questions and discuss this study with anyone at NIH, or with family, friends or your personal physician or other health professional.

# Why is this study being done?

We are investigating an experimental therapy with genetically modified immune cells that target the human papillomavirus (HPV) for vulvar high-grade squamous intraepithelial lesion (HSIL). Vulvar HSIL is caused by infection of the vulva with HPV. In a small percent of patients vulvar HSIL can turn into cancer. The risk of cancer can be reduced by treatment of HSIL. The primary

PATIENT IDENTIFICATION

#### CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

• Adult Patient or

• Parent, for Minor Patient

NIH-2514-1 (07-09) P.A.: 09-25-0099

| CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study |
|---|
| NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |

STUDY NUMBER: 17-C-0116 CONTINUATION:  pages

treatment is surgery to cut out the areas of HSIL. Sometimes a cream that stimulates the immune system may also be used for treatment. Rarely, vulvar HSIL can go away on its own.

Surgery for vulvar HSIL can cause disfigurement or functional impairment. Also, it may not completely remove the disease and may not prevent its recurrence. You may only participate in this study if you have vulvar HSIL that cannot be removed with surgery without causing disfigurement or functional impairment that you would consider unacceptable, or if you have already have had surgery but it failed to control your vulvar HSIL.

This study is being done to determine if a personalized immune treatment can rid the body of HPV infection and thereby cure vulvar HSIL. The immune treatment in this study is called T cell therapy. Immune cells from your blood will be genetically modified in the laboratory to enable them to the HPV infection. The genetically modified cells will then be given back to you through an intravenous infusion similar to a blood transfusion. After the cells are infused you will receive up to two doses of aldesleukin (IL-2) to help the immune cells to survive longer.

In this study we are modifying your immune cells with a retrovirus to give them the ability to attack HPV-16 E6, a protein that is part of HPV. The HPV-16 E6 protein has been found only on cells infected with the HPV virus. We have given immune cells modified with the same genes to other patients. Our laboratory studies show that these cells work much like the cells we have given patients in the past and should be just as safe as those cells, however, we can't predict all of the side effects that may occur.

The purpose of this study is to determine the safe dose of E6 TCR cells in combination with aldesleukin to use in patients who have vulvar HSIL. Although aldesleukin is approved by the Food and Drug Administration (FDA), it is not yet approved by the FDA for patients who have vulvar HSIL. E6 TCR cells are a study treatment not yet approved by the Food and Drug administration.

In a previous clinical trial with E6 TCR T cells, patients had metastatic HPV16+ cancers. A variable number of cells were given. The cell infusions were well-tolerated. Tumor responses occurred in 2 of 12 patients; both responses were at the highest dose of cells. In that trial, patients received chemotherapy prior to cell infusion, which is thought to increase both the clinical activity and the toxicity of the T cells. In the current trial, patients will not receive chemotherapy.

# Why are you being asked to take part in this study?

You are being asked to participate in this study because you have been diagnosed with an HPV-16 associated premalignant condition of the vulva (high-grade squamous intraepithelial lesion (HSIL). In addition, you completed the screening evaluation and were found to be eligible to participate in this research study.

PATIENT IDENTIFICATION

**CONTINUATION SHEET for either:** 

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study |
|---|---|
| | NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |

STUDY NUMBER: 17-C-0116 CONTINUATION:  pages

# How many people will take part in this study?

Up to 18 eligible patients will be enrolled in this study.

# **Description of Research Study**

# The Cell protocol has several stages after screening, which you have already completed:

| Stage | Timeframe | Location | Comments & Instructions |
|---|---|---|---|
| Baseline testing | Occurs over 1-2<br>weeks | Outpatient | Optional vulvar biopsy, photographs of lesion(s), labs, other tests as needed |
| Leukapheresis<br>(see page 4 of<br>this consent<br>document) | Occurs on one day, within 21 days prior to cell infusion | Outpatient | This is a half to full day appointment. |
| Cells and aldesleukin (Day 0) | 1-2 days | Inpatient | Receive the E6 TCR cells IV and then high dose aldesleukin about every 12 hours for up to 2 doses. |
| Recovery | 1-3 days | Inpatient unit | Recover from the effects of treatment. |
| Follow -up | Ongoing for 5 years. | Outpatient | Return to clinic for physical exam, review of side effects, labs |

# What will happen if you take part in this research study?

# Before you begin study therapy

# Work up

Prior to receiving the experimental treatment, you will undergo many tests. These include vulvar biopsies, laboratory tests, and other tests as needed. The vulvar biopsies will be done by a gynecologist. There will be a separate consent for the biopsy.

# **During the study**

#### Cell harvest and growth

You will undergo leukapheresis to obtain your white blood cells. These cells will be grown in the lab and genetically modified to recognize a protein on your precancerous cells. If your cells do not grow, you will not be able to receive the cell infusion. If that happens, we will look at alternative experimental treatments at the NIH Clinical Center or refer you to the care of your referring physician. We usually know after about 4 weeks whether the cells will grow well

| PATIENT IDENTIFICATION | CONTINUATION SHEET for either: |
|---|---|
| | NIH-2514-1 (07-09)<br>NIH-2514-2 (10-84) |
| | P.A.: 09-25-0099 File in Section 4: Protocol Consent |

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study |
|---|---|
| | NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |

STUDY NUMBER: 17-C-0116 CONTINUATION:  pages

enough to be used as an experimental treatment on this protocol. At the time we determine that your cells are not growing, we will inform you and discuss your options with you.

# Leukapheresis

Leukapheresis is a procedure that allows us to remove certain types of blood cells from you and return the rest of your blood. It is a very common procedure that is done routinely here at the NIH with very few risks. During leukapheresis, blood is removed from you through a needle in your arm, circulated through a machine that divides whole blood into red cells, plasma (the serum part), and leukocytes (or white cells), and then the plasma and red cells are returned to you through a second needle in your other arm. If you are receiving the experimental cell therapy, the white blood cells will be used to grow your treatment cells. In addition to the leukapheresis you will undergo as part of your work up, we will also ask you to undergo one additional pheresis procedure between 4 and 6 weeks after your cell treatment to see the impact of this therapy on the immune system and see if cells we gave you are still active.

# Cell Infusion and Aldesleukin Regimen (Day 0 through Day 2)

You will be admitted to the hospital for this procedure. You will be given the cells through an IV (intravenously, or through your veins) over 15 to 30 minutes on day 0. This may be done through a peripheral line (a short tube placed in a vein in your arm), through a "central line," (an IV catheter [or tube] placed in the large vein in your neck or in your chest, or through a PICC line (a peripherally inserted central catheter, which is a thin tube inserted into a vein in your upper arm and is then guided into a large vein in your chest). The doctor will discuss this with you to determine the best method for you. Within 24 hours after your cell infusion you will be given high dose aldesleukin through an IV peripheral line, central line or PICC line. It will be given as a 15-minute infusion about every 12 hours for up to 2 doses. Aldesleukin is a cell growth factor and it is thought that it will help the cells live longer in your body. The day after your cells are infused, we will watch you closely during this entire time for any side effects of this experimental regimen. We will discuss the side effects below and we will include in your care all the medicines and treatments to prevent as many of these side effects as we can and to make you as comfortable as we can.

# When you are finished with the T cell treatment

# Recovery

You will recover in the hospital until you are well enough to go home. This usually takes 1-3 days after you have received cells or your last dose of aldesleukin; however, you may need to stay in the hospital for longer than this before you are well enough to go home. We will continue to give you support medications, do laboratory tests, and watch you closely for any side effects until we feel your condition is stable.

In addition to the laboratory tests to monitor your condition, we will remove between 1 and 9 teaspoons of blood one day after you have received cells, three days after you have received

PATIENT IDENTIFICATION CONTINUATION SHEET for either:

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

MEDICAL RECORD

CONTINUATION SHEET for either:
NIH 2514-1, Consent to Participate in A Clinical Research Study
NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 17-C-0116 CONTINUATION:  pages

cells, then three days per week for one week (Monday, Wednesday, Friday) and then once per week until you are discharged from the hospital to study the effects of this regimen on your immune system. If you experience side effects in your kidneys, we will collect 1 additional teaspoon of blood and about 6 teaspoons of urine to help us determine the cause of these side effects. The maximum amount of blood for research is approximately 2.3 cups in 8 weeks.

### Follow up and Evaluation of Experimental Regimen

We will ask you to return to the NIH Clinical Center frequently for followup visits after you are discharged approximately every month for 3 months. After 3 months, if your lesions have not shrunk, you will be taken off the treatment and you will need to follow up with your physician for care. If your lesions have shrunk after 3 months, you will be seen monthly for another 3 months. If at 6 months, your lesions are still present, you will be taken off the treatment and you will need to follow up with your physician for care. If at 6 months, your tumor has disappeared, you will be seen every three months for two visits, then every 6 months for 2 visits. The follow up visits will probably take about 1 day. At each visit, you will have lab tests and a physical examination. At some of your follow up visits, you may undergo leukapheresis or have about 8 tubes of blood drawn (4 tablespoons) so that we can see the effect this therapy has had on your immune system and if the cells we gave you are still alive. At some followup visits you will have an optional repeat vulvar biopsy (at your 2 week followup, your 1 month followup visit, and at the time you come off-treatment. There will be a separate consent for any biopsies. If you are unwilling or unable to travel to the NIH Clinical Center, we will contact you by phone or e-mail and we may ask you to send us labs and physical exam reports.

After you are taken off treatment, we will contact you once a year for five years to ask you questions about your HSIL, such as whether you have had procedures or other treatments.

#### **Birth Control**

If you are a woman who is breast feeding or pregnant, you may not take part in the study because we don't know how this medicine would affect your baby or your unborn child. If you are a woman who can become pregnant, you will need to practice an effective form of birth control before starting study treatment and for the duration of study participation. If you think that you are pregnant, you should tell your study doctor or nurse at once.

Effective forms of birth control include

- abstinence
- intrauterine device (IUD)
- hormonal [birth control pills, injections, or implants]
- tubal ligation

PATIENT IDENTIFICATION CONTINUATION SHEET for either:

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|
|---|---|

STUDY NUMBER: 17-C-0116 CONTINUATION:  pages

vasectomy of partner(s)

# **Gene Therapy Long Term Follow up (Retroviral Vectors)**

You will be followed on a separate protocol once you are off treatment. There will be a consent process for the separate protocol. Because we do not know the long term side effects of gene therapy, we will ask you to take part in long term follow up for the next 15 years. The Food and Drug Administration (FDA) requires that people who receive gene therapy be watched even after they complete the study. We will ask you questions about your health, and ask you to have a physical exam every year. We will also collect your blood over the next several years. If you return to your referring doctor after treatment here we will ask you to have your doctor send us a copy of your physical exam and your blood samples. We will collect blood samples right after you receive the cells, and at 3, 6 and 12 months after treatment, and then every year after that (2 teaspoons each time). This testing will help us learn if the cells have grown or changed in your body. For this reason, we ask that you continue to provide us with a current address and telephone number, even after you complete this research study.

At the time of your death, no matter the cause, we may request consent from your family for an autopsy. This will allow us to obtain important information about the safety of this experimental treatment. Please discuss this with your family to inform them of this potential request.

# **Risks or Discomforts of Participation**

# What side effects or risks can I expect from being in this study?

The risks and discomforts of this research study can be significant. It is possible, although unlikely, that this experimental treatment may cause your death.

We will discuss the side effects of this experimental treatment with you. You will be given medicines, transfusions, and treatments as needed to prevent or treat the side effects. We will try to make you as comfortable as possible.

#### Leukapheresis

During the leukapheresis procedure, you may have some tingling in your face and lips due to the medicine used to keep your blood from clotting during the procedure. The nurses may give you a calcium-containing antacid to chew that takes away this tingling. Rarely, people may experience lightheadedness or dizziness. We ask that you eat prior to the procedure to prevent this. Rare complications of this procedure are lowered blood pressure, bleeding or bruising where the needles are put in your arms.

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study |
|---|---|
| | NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |

STUDY NUMBER: 17-C-0116 CONTINUATION:  pages

#### **Cell Infusion**

The cells we will be giving you have a type of virus (retrovirus) put into them that makes them able to recognize the HPV E6 protein. Although this retrovirus is not active, there is the rare possibility that it may cause infection. The cells could also cause you to develop another type of cancer, such as leukemia or lymphoma.

#### Potential risks include:

- Fever, chills and shortness of breath, which may last for a few hours (common)
- Lung congestion causing shortness of breath
- Severe reaction to the cells which would include very low blood pressure and damage to your heart, lung, and/or kidneys
- As this is a new experimental therapy which has not been given to patients with your disease, side effects that we do not anticipate that may cause your condition to deteriorate may be encountered. Any new information that becomes available during the course of this study will be shared with you.

# **Medications**

The side effects of high dose aldesleukin and are listed below:

| IL-2 (aldesleukin) side effects | | |
|---|---|---|
| Common (>1 to 10%) | Less common (0.1% to 1%) | Rare (< 0.1%) |
| <ul> <li>Fever, chills, and fatigue</li> <li>Lowered platelet and red blood cell levels that may require transfusions</li> <li>Significant fluid retention causing weight gain (as much as 20 pounds).</li> <li>Low blood pressure</li> <li>Increased heart rate</li> <li>Low urine output</li> </ul> | <ul> <li>Decrease in thyroid function that may require daily thyroid hormone replacement;</li> <li>Abnormal kidney and liver function that can be severe;</li> <li>Abnormal heartbeats or low blood pressure that may require treatment in the ICU.</li> <li>Breathing problems which may need monitoring in ICU and insertion of a</li> </ul> | <ul> <li>Bowel perforation (a hole) requiring longer hospitalization or surgery.</li> <li>Autoimmune disease, where your immune system attacks cells in organs of your body. Should this occur, you will be treated with steroids to stop the immune response.</li> <li>Damage to the heart muscle or heart attack</li> <li>Loss of blood flow to the extremities due to medicines</li> </ul> |
| Swelling in your extremities, | breathing tube. | used to treat very low blood pressure and shock. In one instance a patient had to |

#### PATIENT IDENTIFICATION

#### **CONTINUATION SHEET for either:**

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

MEDICAL RECORD **CONTINUATION SHEET for either:** NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study STUDY NUMBER: 17-C-0116 CONTINUATION:  pages have her lower arm Fluid in your lungs that amputated after treatment can require oxygen with these medicines. Dry mouth, nausea, Aldesleukin is mixed with vomiting and diarrhea; human albumin which could Rash, itching; and cause an allergic reaction or changes in skin or hair potentially transmit viral pigmentation, called infections, although we have vitiligo; not had this occur. Changes in mental status, including confusion, difficulty sleeping or vivid dreams; this can be severe and require sedation and monitoring in the ICU

# **Intravenous Line Placement**

If you require a peripheral IV line, the risks include pain, bleeding, infection and rash/swelling at the insertion site.

If you require a PICC line, it may be inserted under local anesthesia. the risks of the insertion procedure include pain, bleeding, rash/swelling at the insertion site and infection. Long-term risks of a PICC line include infection, a blockage from air that gets into a vein, or a blood clot in the vein. If these occur, it may be necessary to remove the PICC line. These risks will be explained to you in more detail at the time of insertion.

If you require a Central line catheter, it is usually inserted under local anesthesia. The risks associated with the procedure include pain, bleeding, infection, and puncture of the underlying lung. Lung puncture can result in lung collapse, which might require that a chest tube be placed into the chest cavity (usually for a day or two) to help the lung re-inflate. The long-term risks of the catheter include infection and clotting of the vein in which the catheter sits. If these occur, it may be necessary to remove the catheter. These risks will be explained to you in more detail at the time of the insertion.

# Optional vulvar biopsy risks

The risks of a vulvar biopsy include bruising and discomfort at the biopsy site and rarely bleeding and infection.

| PATIENT IDENTIFICATION | CONTINUATION SHEET for either: |
|------------------------|-------------------------------------|
| | NIH-2514-1 (07-09) |
| | NIH-2514-2 (10-84) |
| | P.A.: 09-25-0099 |
| | File in Section 4: Protocol Consent |

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study |
|---|---|
| | NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |

STUDY NUMBER: 17-C-0116 CONTINUATION:  pages

Prior to and throughout this study you will undergo many physical exams to determine the size and extent of your precancer lesion, as well as the impact of the treatment. Multiple blood tests will be performed and some of your serum and lymphocytes will be stored for future testing. Blood and tissue samples collected from you may be stored and used in the future to study scientific questions related to this protocol. If there are any risks to you or your family associated with these future scientific studies which are not covered in this consent form, your consent will be obtained before such studies are performed.

If your disease progresses or recurs after this experimental treatment, then you will no longer receive treatment in this protocol, though you may be eligible to be considered for other protocols at the National Cancer Institute, NIH or referred elsewhere for treatment.

# **Gene Therapy Risk of Cancer and Other Diseases**

We are unsure if this type of gene therapy will cause you to become sick in the future. It is possible that it may cause your immune system or nerves not to work well or cause a sickness of your blood cells or even a cancer (for example leukemia). We do not know if you will develop any of these disorders, but you need to be aware of this possible risk. Children in France and England received gene therapy for a particular disease of the immune system. Most of the children were cured, but 5 children out of 22 later developed leukemia and one died. Experts who looked at these cases thought that the gene therapy caused the leukemia in these children. To watch you for this risk we will be testing your blood as described before.

You will be treated on this gene transfer protocol with a viral vector that was manufactured at the NCI Surgery Branch Vector Production Facility before May 2016. An internal review of the facility that made the vector for this protocol determined that the facility needed to be closed due to manufacturing issues. We know of no additional risks related to the previously produced vector for patients who have received cells with vectors made in this facility as the vectors were extensively tested by outside experts. Therefore, the IRB has determined that the potential benefit to you outweighs the potential risks.

#### **Blood Draws**

Blood will be drawn frequently during your treatment. Most of the blood draws will be to monitor your health during and after the T-cell infusion. In addition, some blood samples will be drawn for research purposes. Additional blood draws might be necessary to investigate T cell responses and serum cytokine levels in cases of clinical events such as rapid regressions of lesions or toxicity. These samples will be used to study how your immune system is affected by the cell therapy. Some of the samples may be used for other or future research conducted by the investigational team or other researchers. Side effects of repeated blood sampling depend in part on how the blood is drawn. If through a central venous catheter, risks include contamination of the catheter which would result in a serious blood stream infection, requiring admission to the hospital and giving you antibiotics through the vein; if blood is drawn through a needle into your

PATIENT IDENTIFICATION

#### **CONTINUATION SHEET for either:**

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|
|---|---|

STUDY NUMBER: 17-C-0116 CONTINUATION:  pages

skin, side-effects could include pain and bruising in the area where the blood was drawn. Other side-effects can include lightheadedness, or rarely, fainting. If you have too much blood taken over a prolonged period, your red blood cell count may drop (this is called "anemia"). As a precaution, we will check your red blood cell level, and give you iron treatment or a blood transfusion if needed.

# **Potential Benefits of Participation**

# Are there benefits to taking part in this study?

The aim of this study is to see if this new experimental treatment will cause your precancerous lesions to go away. The potential benefits could include shrinking of your precancer or lessening of your symptoms, such as pain, that are caused by the lesions. Because there is no information about the E6 TCR therapy effect on your type of precancer, we do not know if you will personally benefit from taking part in this study, although the knowledge gained from this study may benefit others in the future who have this precancer.

# **Alternative Approaches or Treatments**

# What other choices do I have if I do not take part in this study?

Instead of being in this study, you have these options:

- Getting treatment or care for your precancer without being in a study, such as surgery to remove the lesion(s). This is called *surgical excision*. Another treatment option for some individuals is topical imiquimod, a cream that is applied directly to the lesions.
- Taking part in another study

Please talk to your doctor about these and other options.

# **Stopping Therapy**

Your doctor may decide to stop your therapy for the following reasons:

- if he/she believes that it is in your best interest
- if you become pregnant
- if your disease comes back during treatment
- if you have side effects from the treatment that your doctor thinks are too severe
- if new information shows that another treatment would be better for you

In this case, you will be informed of the reason therapy is being stopped.

# PATIENT IDENTIFICATION CONTINUATION SHEET for either: NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099 File in Section 4: Protocol Consent

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|
|---|---|

STUDY NUMBER: 17-C-0116 CONTINUATION:  pages

You can stop taking part in the study at any time. However, if you decide to stop taking part in the study, we would like you to talk to the study doctor and your regular doctor first.

If you decide at any time to withdraw your consent to participate in the trial, we will not collect any additional medical information about you. However, according to FDA guidelines, information collected on you up to that point may still be provided to sponsor. If you withdraw your consent and leave the trial, any samples of yours that have been obtained for the study and stored at the NCI can be destroyed upon request. However, any samples and data generated from the samples that have already been distributed to other researchers or placed in the research databases can**not** be recalled and destroyed.

# Research Subject's Rights

#### What are the costs of taking part in this study?

If you choose to take part in the study, the following will apply, in keeping with the NIH policy:

- You will receive study treatment at no charge to you. This may include surgery, medicines, laboratory testing, x-rays or scans done at the Clinical Center, National Institutes of Health (NIH), or arranged for you by the research team to be done outside the Clinical Center, NIH if the study related treatment is not available at the NIH.
- There are limited funds available to cover the cost of some tests and procedures performed outside the Clinical Center, NIH. You may have to pay for these costs if they are not covered by your insurance company.
- Medicines that are not part of the study treatment will not be provided or paid for by the Clinical Center, NIH.
- Once you have completed taking part in the study, medical care will no longer be provided by the Clinical Center, NIH.

#### Will your medical information be kept private?

We will do our best to make sure that the personal information in your medical record will be kept private. However, we cannot guarantee total privacy. Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- The National Cancer Institute (NCI) and other government agencies, like the Food and Drug Administration (FDA), which are involved in keeping research safe for people.
- National Cancer Institute Institutional Review Board

PATIENT IDENTIFICATION CONTINUATION SHEET for either:

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|
| STUDY NUMBER: 17-C-0116 | CONTINUATION: pages |

• The study Sponsor (Center for Cancer Research)

• Qualified representatives from Kite Pharma, the pharmaceutical company who is a collaborator in the production of the E6 TCR T cells.

A description of this clinical trial will be available on <a href="http://www.Clinicaltrials.gov">http://www.Clinicaltrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most the Web site will include a summary of the results. You can search this Web site at any time.

#### **Conflict of Interest**

The National Institutes of Health (NIH) reviews NIH staff researchers at least yearly for conflicts of interest. This process is detailed in a Protocol Review Guide. You may ask your research team for a copy of the Protocol Review Guide or for more information. Members of the research team who do not work for the NIH are expected to follow these guidelines but they do not need to report their personal finances to the NIH.

Members of the research team working on this study may have up to \$15,000 of stock in the companies that make products used in this study. This is allowed under federal rules and is not a conflict of interest.

The National Institutes of Health and the research team for this study have developed the E6 TCR treatment being used in this study. This means it is possible that the results of this study could lead to payments to NIH scientists and to the NIH. By law, government scientists are required to receive such payments for their inventions. You will not receive any money from the development of the E6 TCR therapy.

The National Institutes of Health and the research team for this study are using the E6 TCR developed by Kite Pharma through a joint study with your researchers and the company. The company also provides financial support for this study.

#### **Use of Specimens and Data for Future Research**

To advance science, it is helpful for researchers to share information they get from studying human samples. They do this by putting it into one or more scientific databases, where it is stored along with information from other studies. A researcher who wants to study the information must apply to the database and be approved. Researchers use specimens and data stored in scientific databases to advance science and learn about health and disease.

We plan to keep some of your specimens and data that we collect and use them for future research and share them with other researchers. We will not contact you to ask about each of these future uses. These specimens and data will be stripped of identifiers such as name, address or account number, so that they may be used for future research on any topic and shared broadly for research purposes. Your specimens and data will be used for research purposes only and will

PATIENT IDENTIFICATION CONTINUATION SHEET for either:

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|
|---|---|

STUDY NUMBER: 17-C-0116 CONTINUATION:  pages

not benefit you. It is also possible that the stored specimens and data may never be used. Results of research done on your specimens and data will not be available to you or your doctor. It might help people who have cancer and other diseases in the future.

If you do not want your stored specimens and data used for future research, please contact us in writing and let us know that you do not want us to use your specimens and/or data. Then any specimens that have not already been used or shared will be destroyed and your data will not be used for future research. However, it may not be possible to withdraw or delete materials or data once they have been shared with other researchers.

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

#### MEDICAL RECORD

#### CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

Adult Patient or

• Parent, for Minor Patient

STUDY NUMBER: 17-C-0116

CONTINUATION:  pages

# OTHER PERTINENT INFORMATION

1. Confidentiality. When results of an NIH research study are reported in medical journals or at scientific meetings, the people who take part are not named and identified. In most cases, the NIH will not release any information about your research involvement without your written permission. However, if you sign a release of information form, for example, for an insurance company, the NIH will give the insurance company information from your medical record. This information might affect (either favorably or unfavorably) the willingness of the insurance company to sell you insurance.

The Federal Privacy Act protects the confidentiality of your NIH medical records. However, you should know that the Act allows release of some information from your medical record without your permission, for example, if it is required by the Food and Drug Administration (FDA), members of Congress, law enforcement officials, or authorized hospital accreditation organizations.

- 2. Policy Regarding Research-Related Injuries. The Clinical Center will provide short-term medical care for any injury resulting from your participation in research here. In general, no long-term medical care or financial compensation for research-related injuries will be provided by the National Institutes of Health, the Clinical Center, or the Federal Government. However, you have the right to pursue legal remedy if you believe that your injury justifies such action.
- 3. Payments. The amount of payment to research volunteers is guided by the National Institutes of Health policies. In general, patients are not paid for taking part in research studies at the National Institutes of Health. Reimbursement of travel and subsistence will be offered consistent with NIH guidelines.
- **4. Problems or Questions.** If you have any problems or questions about this study, or about your rights as a research participant, or about any research-related injury, contact the Principal Investigator, Christian S. Hinrichs, M.D., Building 10, Room 4B04, Telephone: 240-760-6059. You may also call the Clinical Center Patient Representative at 301-496-2626 or the Office of the Clinical Director at 240-760-6070.
- **5. Consent Document.** Please keep a copy of this document in case you want to read it again.

PATIENT IDENTIFICATION

# CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY (Continuation Sheet)

• Adult Patient or

• Parent, for Minor Patient

NIH-2514-1 (07-09) P.A.: 09-25-0099

MEDICAL RECORD

# CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

Adult Patient or

• Parent, for Minor Patient

STUDY NUMBER: 17-C-0116

CONTINUATION:  pages

| COMPLETE APPROPRIATE ITEM(S) BELOW: | | | |
|---|---|---|---|
| A. Adult Patient's Consent | | B. Parent's Permission for Minor Patient. | |
| I have read the explanation about this study<br>and have been given the opportunity to discuss<br>it and to ask questions. I hereby consent to<br>take part in this study. | | I have read the explanation about this study<br>and have been given the opportunity to discuss<br>it and to ask questions. I hereby give<br>permission for my child to take part in this<br>study. | |
| | | (Attach NIH 2514-2, Minor's Asso<br>applicable.) | ent, if |
| Signature of Adult Patient/ Legal Representative | Date | Signature of Parent(s)/ Guardian | Date |
| Print Name | | Print Name | |
| C. Child's Verbal Assent (If App | licable) | | |
| The information in the above conserparticipate in the study. | nt was descri | bed to my child and my child agree | s to |
| Signature of Parent(s)/Guardian | Date | Print Name | |
| THIS CONSENT DOCUMENT HAS BEEN APPROVED FOR USE FROM SEPTEMBER 24, 2018 THROUGH APRIL 8, 2019. | | | |
| Signature of Investigator | Date | Signature of Witness | Date |
| Print Name | | Print Name | |

PATIENT IDENTIFICATION

# **CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY (Continuation Sheet)**

• Adult Patient or

• Parent, for Minor Patient

NIH-2514-1 (07-09) P.A.: 09-25-0099